CLINICAL TRIAL: NCT00273052
Title: A Randomized, Double-Blind, Multi-Center Study Comparing the Effects of Carvedilol Phosphate Modified Release Formulation (COREG- MR) With Metoprolol Succinate (TOPROL XL) on the Lipid Profile in Normolipidemic, or Mildly Dyslipidemic Hypertensive Patients
Brief Title: COREG MR Versus TOPROL-XL On The Lipid Profile Of Normolipidemic Or Mildly Dyslipidemic Patients With Hypertension
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: COR103561
Record Dates: First submitted 2006-01-05; First posted 2006-01-09 (Estimated); Results first posted 2010-02-01 (Estimated); Last update posted 2018-06-25 (Actual); Status verified 2018-03

CONDITIONS: Hypertension
Keywords: hypertension
MeSH Terms: conditions — Hypertension | interventions — Metoprolol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Carvedilol Phosphate modified release formulation (Experimental)
  Interventions: Drug: Carvedilol Phosphate modified release formulation
- metoprolol succinate (Active Comparator)
  Interventions: Drug: metoprolol succinate

INTERVENTIONS:
Drug: Carvedilol Phosphate modified release formulation
  Arms: Carvedilol Phosphate modified release formulation
Drug: metoprolol succinate
  Other Names: Carvedilol Phosphate modified release formulation
  Arms: metoprolol succinate

SUMMARY:
This study was designed to determine whether treatment with COREG MR is more effective at maintaining a better lipid profile than treatment with TOPROL-XL for hypertension.

ELIGIBILITY:
Inclusion Criteria:

* Documented history of hypertension
* Triglycerides of 120-400 mg/mL
* LDLc levels not requiring lipid lowering medication.

Exclusion Criteria:

* Has known contraindication to alpha- or beta-blocker therapy.
* Has taken any non-ocular beta-blockers within three months before screening.
* Has Type I or II diabetes.
* Taking lipid lowering medications.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 514 (Actual)
Dates: Start 2006-01-05; Primary Completion 2007-12-01 (Actual); Study Completion 2007-12-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (103):
- United States (87):
  - GSK Investigational Site, Birmingham, Alabama
  - GSK Investigational Site, Montgomery, Alabama
  - GSK Investigational Site, Chandler, Arizona
  - GSK Investigational Site, Mesa, Arizona
  - GSK Investigational Site, Phoenix, Arizona
  - GSK Investigational Site, Tucson, Arizona
  - GSK Investigational Site, Fayetteville, Arkansas
  - GSK Investigational Site, Little Rock, Arkansas
  - GSK Investigational Site, Carmichael, California
  - GSK Investigational Site, Healdsburg, California
  - GSK Investigational Site, Irvine, California
  - GSK Investigational Site, La Jolla, California
  - GSK Investigational Site, Los Angeles, California
  - GSK Investigational Site, Mission Viejo, California
  - GSK Investigational Site, Poway, California
  - GSK Investigational Site, Sacramento, California
  - GSK Investigational Site, San Diego, California
  - GSK Investigational Site, Spring Valley, California
  - GSK Investigational Site, Stockton, California
  - GSK Investigational Site, Torrance, California
  - GSK Investigational Site, Vista, California
  - GSK Investigational Site, Avon, Connecticut
  - GSK Investigational Site, Altamonte Springs, Florida
  - GSK Investigational Site, Clearwater, Florida
  - GSK Investigational Site, Fort Lauderdale, Florida
  - GSK Investigational Site, Jacksonville, Florida
  - GSK Investigational Site, Pembroke Pines, Florida
  - GSK Investigational Site, Atlanta, Georgia
  - GSK Investigational Site, Marietta, Georgia
  - GSK Investigational Site, Roswell, Georgia
  - GSK Investigational Site, Aurora, Illinois
  - GSK Investigational Site, Chicago, Illinois
  - GSK Investigational Site, Gillespie, Illinois
  - GSK Investigational Site, Vernon Hills, Illinois
  - GSK Investigational Site, Evansville, Indiana
  - GSK Investigational Site, Indianapolis, Indiana
  - GSK Investigational Site, Wichita, Kansas
  - GSK Investigational Site, Bossier City, Louisiana
  - GSK Investigational Site, Auburn, Maine
  - GSK Investigational Site, Natick, Massachusetts
  - GSK Investigational Site, Taunton, Massachusetts
  - GSK Investigational Site, West Yarmouth, Massachusetts
  - GSK Investigational Site, Detroit, Michigan
  - GSK Investigational Site, Brooklyn Center, Minnesota
  - GSK Investigational Site, Olive Branch, Mississippi
  - GSK Investigational Site, Springfield, Missouri
  - GSK Investigational Site, St Louis, Missouri
  - GSK Investigational Site, Omaha, Nebraska
  - GSK Investigational Site, Henderson, Nevada
  - GSK Investigational Site, Las Vegas, Nevada
  - GSK Investigational Site, Brick, New Jersey
  - GSK Investigational Site, Elizabeth, New Jersey
  - GSK Investigational Site, Albuquerque, New Mexico
  - GSK Investigational Site, East Syracuse, New York
  - GSK Investigational Site, Endwell, New York
  - GSK Investigational Site, Fishkill, New York
  - GSK Investigational Site, New York, New York
  - GSK Investigational Site, Charlotte, North Carolina
  - GSK Investigational Site, Raleigh, North Carolina
  - GSK Investigational Site, Statesville, North Carolina
  - GSK Investigational Site, Wilmington, North Carolina
  - GSK Investigational Site, Winston-Salem, North Carolina
  - GSK Investigational Site, Cincinnati, Ohio
  - GSK Investigational Site, Cleveland, Ohio
  - GSK Investigational Site, Kettering, Ohio
  - GSK Investigational Site, Oklahoma City, Oklahoma
  - GSK Investigational Site, Erie, Pennsylvania
  - GSK Investigational Site, Warminster, Pennsylvania
  - GSK Investigational Site, West Chester, Pennsylvania
  - GSK Investigational Site, Columbia, South Carolina
  - GSK Investigational Site, Greer, South Carolina
  - GSK Investigational Site, Hartsville, South Carolina
  - GSK Investigational Site, Simpsonville, South Carolina
  - GSK Investigational Site, Bristol, Tennessee
  - GSK Investigational Site, Kingsport, Tennessee
  - GSK Investigational Site, Corpus Christi, Texas
  - GSK Investigational Site, San Antonio, Texas
  - GSK Investigational Site, Salt Lake City, Utah
  - GSK Investigational Site, Burke, Virginia
  - GSK Investigational Site, Galax, Virginia
  - GSK Investigational Site, Manassas, Virginia
  - GSK Investigational Site, Newport News, Virginia
  - GSK Investigational Site, Richmond, Virginia
  - GSK Investigational Site, Springfield, Virginia
  - GSK Investigational Site, Virginia Beach, Virginia
  - GSK Investigational Site, Walla Walla, Washington
  - GSK Investigational Site, Lewisburg, West Virginia
- Canada (13):
  - GSK Investigational Site, Calgary, Alberta
  - GSK Investigational Site, Edmonton, Alberta
  - GSK Investigational Site, St. John's, Newfoundland and Labrador
  - GSK Investigational Site, Truro, Nova Scotia
  - GSK Investigational Site, Brampton, Ontario
  - GSK Investigational Site, Greater Sudbury, Ontario
  - GSK Investigational Site, London, Ontario
  - GSK Investigational Site, Newmarket, Ontario
  - GSK Investigational Site, Peterborough, Ontario
  - GSK Investigational Site, Sarnia, Ontario
  - GSK Investigational Site, Gatineau, Quebec
  - GSK Investigational Site, Mirabel, Quebec
  - GSK Investigational Site, Trois-Rivières, Quebec
- Puerto Rico (3):
  - GSK Investigational Site, Ponce
  - GSK Investigational Site, Rio Piedras
  - GSK Investigational Site, Río Grande

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Statistical Analysis Plan: COR103561 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: COR103561 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: COR103561 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: COR103561 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: COR103561 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: COR103561 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: COR103561 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Groups:
- Coreg CR: Carvedilol Phosphate Extended Release 20 mg, 40 mg, and 80 mg Capsules QD (once daily)
- Toprol XL: Metoprolol Succinate Extended Release 50 mg, 100 mg, and 200 mg Tablets QD (once daily)
Period: Overall Study
Arm/Group | Coreg CR | Toprol XL
Started | 290 | 278
Completed | 221 | 190
Not Completed | 69 | 88
Not completed — Withdrawal by Subject | 16 | 19
Not completed — Adverse Event | 21 | 19
Not completed — Protocol Violation | 14 | 18
Not completed — Lost to Follow-up | 7 | 25
Not completed — Lack of Efficacy | 6 | 4
Not completed — Non-Compliance | 3 | 1
Not completed — Other | 2 | 0
Not completed — Worsening serum lipid levels | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Coreg CR | Toprol XL | Total
Number analyzed (Participants) | 290 | 278 | 568
Age, Customized [Number; unit: participants]
  < 65 years | 260 | 244 | 504
  >=65 years | 30 | 34 | 64
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 137 | 133 | 270
  Male | 153 | 145 | 298
Race/Ethnicity, Customized [Number; unit: participants]
  Black | 24 | 28 | 52
  White/Caucasian | 239 | 226 | 465
  Other | 27 | 24 | 51

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Triglycerides Levels by Treatment Group at Maintenance Month 6
Description: Blood draw for triglyceride levels. Full beta quantification test performed which uses ultracentrifugation to partially separate lipoprotein classes and is the basis for the reference methods. Change = Month 6 value minus Baseline value.
Time Frame: Baseline and Month 6
Population: The Intent to Treat (ITT-E) Population was used for analysis of the efficacy results and consisted of all subjects who randomized, received at least one dose of study medication, and had both a baseline and at least one on-therapy value for an efficacy parameter during the maintenance phase(number of participants will vary between measures).
Measure: Number; unit: mg/dL
Arm/Group | Coreg CR | Toprol XL
Number analyzed (Participants) | 235 | 206
mg/dL | 2.65 | 10.39
Statistical Analysis 1: Comparison: Coreg CR vs Toprol XL; Test type: Superiority or Other; p = 0.0141, ANCOVA; Median Difference (Net) = -8.026, 95% CI [-15.35 to -0.67] — Median difference = Coreg CR - Toprol XL

2. Primary Outcome: Change From Baseline in High-Density Lipoprotein Cholesterol (HDL-C) Levels by Treatment Group at Maintenance Month 6
Description: Blood draw for HDL-C levels. Full beta Quant test performed with HDL subclasses. Change = Month 6 value minus Baseline value.
Time Frame: Baseline and Month 6
Population: as for outcome 1
Measure: Number; unit: mg/dL
Arm/Group | Coreg CR | Toprol XL
Number analyzed (Participants) | 235 | 206
mg/dL | -4.4 | -5.1
Statistical Analysis 1: Comparison: Coreg CR vs Toprol XL; Test type: Superiority or Other; p = 0.6068, ANCOVA; Mean Difference (Net) = 0.7, 95% CI [-2.4 to 3.9] — Mean difference = Coreg CR - Toprol XL

3. Secondary Outcome: Change From Baseline in Log Transformed High Sensitivity C-reactive Protein (Hs-CRP) by Treatment Group at Maintenance Month 6
Description: Blood draw for hs-CRP. Change = Month 6 value minus Baseline value.
Time Frame: Baseline and Month 6
Population: as for outcome 1
Measure: Number; unit: mg/dL
Arm/Group | Coreg CR | Toprol XL
Number analyzed (Participants) | 231 | 203
mg/dL | -1.76 | 0.49

4. Secondary Outcome: Change From Baseline in Log Transformed Lipoprotein-associated Phospholipase A2 (LpPLA2) by Treatment Group at Maintenance Month 6
Description: Blood draw for LpPLA2 activity. Change = Month 6 value minus Baseline value.
Time Frame: Baseline and Month 6
Population: as for outcome 1
Measure: Number; unit: mcmol/min/L
Arm/Group | Coreg CR | Toprol XL
Number analyzed (Participants) | 222 | 189
mcmol/min/L | -2.38 | -2.23

5. Secondary Outcome: Change From Baseline in Blood Pressure by Treatment Group at Maintenance Month 6
Description: Manual physical examination (cuff blood pressure). Change = Month 6 value minus Baseline value.
Time Frame: Baseline and Month 6
Population: as for outcome 1
Measure: Number; unit: mm Hg
Arm/Group | Coreg CR | Toprol XL
Number analyzed (Participants) | 280 | 269
mm Hg
  Systolic Blood Pressure | -15.90 | -16.23
  Diastolic Blood Pressure | -10.89 | -11.06

6. Secondary Outcome: Change From Baseline in Heart Rate by Treatment Group at Maintenance Month 6
Description: Manual physical examination. Change = Month 6 value minus Baseline value. (BPM=beats per minute)
Time Frame: Baseline and Month 6
Population: as for outcome 1
Measure: Number; unit: bpm
Arm/Group | Coreg CR | Toprol XL
Number analyzed (Participants) | 280 | 269
bpm | -5.98 | -6.07

7. Secondary Outcome: Change From Baseline in Weight by Treatment Group at Maintenance Month
Description: Manual physical examination. Change = Month 6 value minus Baseline value.
Time Frame: Baseline and Month 6
Population: as for outcome 1
Measure: Number; unit: kg
Arm/Group | Coreg CR | Toprol XL
Number analyzed (Participants) | 280 | 269
kg | 1.01 | 0.73

8. Secondary Outcome: Change From Baseline in Additional Lipid Parameters by Treatment Group With Unit of Measures of mg/dL at Maintenance Month 6
Description: Blood draw for lipid levels. Full beta Quant test performed with HDL subclasses and IDL. IDL=Intermediate density lipoproteins, LDL=Low-density lipoprotein, VLDL=Very Low density lipoprotein, HDL=High-density lipoprotein. Change = Month 6 value minus Baseline value.
Time Frame: Baseline and Month 6
Population: as for outcome 1
Measure: Number; unit: mg/dL
Arm/Group | Coreg CR | Toprol XL
Number analyzed (Participants) | 280 | 269
mg/dL
  Total Serum Cholesterol | 0.1 | -0.7
  Low-Density Lipoprotein (LDL) | -1.1 | -1.7
  Low+Very Low Density Lipoprotein | 0.9 | 0.4
  High-Density Lipoprotein 2 (HDL2) | -1.45 | -6.5
  High-Density Lipoprotein 3 (HDL3) | -4.0 | -3.5
  Low-Density Lipoprotein-Relative Flotation | 0.166 | -1.360
  Intermediate Density Lipoproteins+VLDL | 2.0 | 5.6

9. Secondary Outcome: Change From Baseline in Additional Lipid Parameters by Treatment Group With Unit of Measures of g/L at Maintenance Month 6
Description: Blood draw for lipid levels. Full beta Quant test performed. Change = Month 6 value minus Baseline value.
Time Frame: Baseline and Month 6
Population: as for outcome 1
Measure: Number; unit: g/L
Arm/Group | Coreg CR | Toprol XL
Number analyzed (Participants) | 280 | 269
g/L
  Apolipoprotein A-1 (Apo-A1) | -1.82 | -3.45
  Apolipoprotein B (Apo-B) | -1.16 | 0.81

10. Secondary Outcome: Change From Baseline in Fasting Insulin (Glycemic Parameter) by Treatment Group at Maintenance Month 6
Description: Blood draw for glycemia levels. Full beta Quant test performed. Test for Fasting plasma glucose, HbA1c, fasting insulin. Homeostasis model Assessment (HOMA) is a computer-generated model consisting of non-linear empirical equations solved numerically to predict glucose, Insulin and C-peptide concentrations in fasting subjects for insulin sensitivity (%S). Change = Month 6 value minus Baseline value.
Time Frame: Baseline and Month 6
Population: as for outcome 1
Measure: Number; unit: uIU/mL
Arm/Group | Coreg CR | Toprol XL
Number analyzed (Participants) | 280 | 269
uIU/mL | -1.21 | 1.35

11. Secondary Outcome: Change From Baseline in Hemoglobin A1c (HbA1c) (Glycemic Parameter) by Treatment Group at Maintenance Month 6
Description: as for outcome 10
Time Frame: Baseline and Month 6
Population: as for outcome 1
Measure: Number; unit: Percent Change
Arm/Group | Coreg CR | Toprol XL
Number analyzed (Participants) | 280 | 269
Percent Change | 0.01 | 0.04

12. Secondary Outcome: Change From Baseline in c-Peptide (Glycemic Parameter) by Treatment Group at Maintenance Month 6
Description: as for outcome 10
Time Frame: Baseline and Month 6
Population: as for outcome 1
Measure: Number; unit: ng/mL
Arm/Group | Coreg CR | Toprol XL
Number analyzed (Participants) | 280 | 269
ng/mL | -0.23 | 0.20

13. Secondary Outcome: Change From Baseline in Homeostasis Model Assessment (Glycemic Parameter) by Treatment Group at Maintenance Month 6
Description: as for outcome 10
Time Frame: Baseline and Month 6
Population: as for outcome 1
Measure: Number; unit: Percent Change
Arm/Group | Coreg CR | Toprol XL
Number analyzed (Participants) | 280 | 269
Percent Change | 2.05 | -4.14

14. Secondary Outcome: Change From Baseline in Fasting Plasma Glucose (FPG) (Glycemic Parameter) by Treatment Group at Maintenance Month 6
Description: as for outcome 10
Time Frame: Baseline and Month 6
Population: as for outcome 1
Measure: Number; unit: mg/dL
Arm/Group | Coreg CR | Toprol XL
Number analyzed (Participants) | 280 | 269
mg/dL | 0.94 | 1.20

ADVERSE EVENTS:
Groups:
- Coreg CR; Toprol XL: Results include only treatment emergent events.
Arm/Group | Coreg CR | Toprol XL
Serious Adverse Events (participants affected / at risk) | 8 | 5
Other Adverse Events (participants affected / at risk) | 186 | 160
SERIOUS ADVERSE EVENTS; cells are participants affected / at risk:
Term (organ system) | Coreg CR | Toprol XL
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/290 | 1/278
Chest discomfort (General disorders) | 1/290 | 0/278
Colitis ischaemic (Gastrointestinal disorders) | 1/290 | 0/278
Depression suicidal (Psychiatric disorders) | 1/290 | 0/278
Gastroesophagael reflux disease (Gastrointestinal disorders) | 1/290 | 0/278
Hydronephrosis (Renal and urinary disorders) | 0/290 | 1/278
Hypertension (Vascular disorders) | 1/290 | 0/278
Myocardial Infarction (Cardiac disorders) | 1/290 | 0/278
Orthostatic hypotension (Nervous system disorders) | 0/290 | 1/278
Palpitations (Cardiac disorders) | 1/290 | 0/278
Peridiverticular abscess (Infections and infestations) | 0/290 | 1/278
Presyncope (Nervous system disorders) | 0/290 | 1/278
Umbilical hernia (Gastrointestinal disorders) | 1/290 | 0/278
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected / at risk:
Term (organ system) | Coreg CR | Toprol XL
Headache (Nervous system disorders) | 42/290 | 33/278
Edema Peripheral (General disorders) | 29/290 | 25/278
Fatigue (General disorders) | 22/290 | 29/278
Dizziness (Nervous system disorders) | 28/290 | 18/278
Nasopharyngitis (Infections and infestations) | 16/290 | 17/278
Upper Respiratory Tract Infection (Infections and infestations) | 19/290 | 12/278
Nausea (Gastrointestinal disorders) | 18/290 | 11/278
Diarrhea (Gastrointestinal disorders) | 12/290 | 15/278

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centres of a multi-centre trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.